CLINICAL TRIAL: NCT06607146
Title: Assessing the Effect of Computer-based Auditory Training on Adult Cochlear Implant Speech and Quality-of-life Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew L. Carlson, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-010096
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cochlear Implants; Bilateral Sensorineural Hearing Loss
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator)
  Interventions: Behavioral: Standard of Care
- Experimental Group (Experimental)
  Interventions: Behavioral: Sound Success

INTERVENTIONS:
Behavioral: Sound Success — Subjects will be instructed to perform auditory training with the Sound Success computer-based auditory training program. This is a free program that requires a brief account registration. Subjects will be instructed to perform auditory training on a personal device and will be recommended a target usage of at least 30 minutes 5 times per week.
  Arms: Experimental Group
Behavioral: Standard of Care — Subjects will be provided a list of common exercises for auditory training. This is the current standard of care at our institution.
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare the effectiveness of a free computer-based auditory training program, Sound Success (Advanced Bionics, Valencia, CA), with the current standard of care of patient-directed auditory training in improving common measures of speech recognition and cochlear implant (CI) specific quality-of-life in new adult CI recipients in their first year post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of bilateral moderate-to-profound sensorineural hearing loss who are undergoing unilateral or simultaneous bilateral cochlear implantation at the Mayo Clinic in Rochester MN.

Exclusion Criteria:

* Patients undergoing revision implantation, completion bilateral cochlear implantation, or implantation for unilateral deafness will be excluded from enrollment
* Patients unable or unwilling to use a computer or similar device will be excluded from enrollment.
* Patients will be excluded if they speak a language not supported by the Sound Success platform. Sound Success is available in English, Spanish, French, Italian, Dutch, Polish, and Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cochlear Implant Quality of Life-35 Profile | Baseline, 3 months, 6 months, 12 months
  The Cochlear Implant Quality of Life-35 (CIQOL-35) Profile is a patient reported questiornaire that assesses the functional abilities of adult cochlear implant recipients within 6 domains: communication, assessing communication ability in different circumstances; emotional, assessing the impact of hearing on emotional well-being; entertainment, assessing the ability to enjoy television, radio, and music; environmental, assessing the ability to distinguish and localize environmental sounds; listening effort, assessing effort and fatigue associated with receptive communication; and social, assessing the ability to interact and enjoy interaction with groups. Scores are calculated for each domain and ranged from 0 (poorest Quality of Life) to 100 (highest Quality of Life).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Carlson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States